CLINICAL TRIAL: NCT00493103
Title: Congenital Hypothyroidism Due to Thyroglobulin Mutations in an Inbred Brazilian Family: A Novel Compound Heterozygous Constellation and Intronic Mutation Related to Fetal Goiter.
Brief Title: TG Gene Mutations and Congenital Hypothyroidism
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Other Study IDs: PRN989/03
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Congenital Hypothyroidism
Keywords: thyroglobulin gene; congenital hypothyroidism; gene mutations; fetal goiter; iodine nutrition
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to identify mutations in the thyroglobulin gene that might be present in patients with fetal goiter and congenital goiter hypothyroidism.

DETAILED DESCRIPTION:
Congenital goitrous hypothyroid is commonly linked to thyroglobulin (TG) gene mutations.We aim to identify mutations in the TG gene that might be present in patients with fetal goiter and congenital goiter hypothyroidism.Four related patients with congenital goiter hypothyroidism from an inbred family were studied.Recombinant human TSH stimulation test, DNA sequencing and protein computer analysis were performed.We identified a novel compound heterozygous constellation (IVS30+1G>T/A2215D) in two siblings. It was also identified a homozygous intronic mutation (IVS30+1G>T) in their cousins, one of them with fetal goiter. The mutation IVS30+1G>T promotes an aberrant splicing and loss of the entire exon 30 (138 nt) in the resulting messenger RNA. The recent described mutation A2215D is located in the ACHE-like domain, which functions as a dimerization domain, facilitating efficient intracellular transport of the protein. Protein computer analysis suggested that the A2215D mutation causes TG structural alterations.A novel compound heterozygous constellation (IVS30+1G>T/A2215D) and the previously described mutation (IVS30+1G>T) that cause severe congenital hypothyroidism due to defective TG synthesis have been identified. The mutation IVS30+1G>T may be related to fetal goiter and hypothyroidism due to TG instability and impaired TG export to the colloid. This study shows the efficiency of the use of rhTSH in the differential diagnosis of CH due to TG defective synthesis and the importance of molecular diagnosis of CH for possible intrauterine treatment, thereby avoiding damage to the neuropsychomotor system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital hypothyroidism due to thyroglobulin defective synthesis.

Exclusion Criteria:

* Patients with another disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-07; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Pardo, Principal Investigator — University of Sao Paulo; Geraldo Medeiros-Neto, Study Director — University of Sao Paulo